CLINICAL TRIAL: NCT04120194
Title: A Phase 3, Randomized, Observer-blinded, Active-controlled Trial to Evaluate Immunogenicity & Safety of a Recombinant Quadrivalent Nanoparticle Influenza Vaccine (Quad-NIV) With Matrix-M1™ Adjuvant Against Fluzone® Quadrivalent in Clinically Stable Adults ≥ 65 Years of Age
Brief Title: Phase 3 Pivotal Trial of NanoFlu™ in Older Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: qNIV-E-301
Record Dates: First submitted 2019-10-07; First posted 2019-10-09 (Actual); Results first posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NanoFlu (Experimental): NanoFlu will be administered as a single dose (0.5 mL) in the arm muscle on Day 0.
  Interventions: Biological: NanoFlu
- Fluzone Quadrivalent (Active Comparator): Fluzone Quadrivalent will be administered as a single dose (0.5 mL) in the arm muscle on Day 0.
  Interventions: Biological: Fluzone Quadrivalent

INTERVENTIONS:
Biological: NanoFlu — Investigational quadrivalent seasonal influenza vaccine for the 2019-20 Northern hemisphere influenza season.
  Other Names: Quad-NIV
  Arms: NanoFlu
Biological: Fluzone Quadrivalent — Licensed quadrivalent seasonal influenza vaccine for the 2019-20 Northern hemisphere influenza season.
  Arms: Fluzone Quadrivalent

SUMMARY:
A Phase 3, randomized, observer-blinded, active-controlled trial to evaluate the immunogenicity and safety of a recombinant quadrivalent nanoparticle influenza vaccine with Matrix-M1 adjuvant (NanoFlu) compared with a licensed quadrivalent inactivated influenza vaccine in adults ≥ 65 years of age. Both vaccines were formulated with the 4 influenza strains recommended for the 2019-20 Northern hemisphere influenza season. 2654 subjects were enrolled and randomized into 1 of 2 treatment groups to receive either NanoFlu or active comparator. Subjects were followed for approximately 1 year following injection; with primary immunogenicity analyses based on Day 28 sera. This trial was conducted in the United States at approximately 19 clinical sites.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically-stable adult male or female, ≥ 65 years of age. Subjects may have 1 or more chronic medical diagnoses, but should be clinically stable as assessed by:

   * Ambulatory status, living independently in the community or in a residential facility providing minimal assistance (eg, meal preparation and transport),
   * Absence of changes in medical therapy within 1 month due to treatment failure or toxicity,
   * Absence of medical events qualifying as serious adverse events within the prior 2 months, and
   * Absence of known, current, and life-limiting diagnoses which render survival to completion of the protocol unlikely in the opinion of the investigator.
2. Willing and able to give informed consent prior to trial enrollment, and
3. Living in the community and able to attend trial visits, comply with trial requirements, and provide timely, reliable, and complete reports of adverse events.

Exclusion Criteria:

1. Participation in research involving investigational product (drug / biologic / device) within 45 days before planned date of study vaccination.
2. Participation in any previous Novavax influenza vaccine clinical trial(s).
3. History of a serious reaction to prior influenza vaccination, known allergy to constituents of Fluzone Quadrivalent or polysorbate 80.
4. History of Guillain-Barré Syndrome (GBS) within 6 weeks following a previous influenza vaccine.
5. Received any vaccine in the 4 weeks preceding the trial vaccination and any influenza vaccine within 6 months preceding the trial vaccination.
6. Any known or suspected immunosuppressive illness, congenital or acquired, based on medical history and/or physical examination.
7. Chronic administration (defined as more than 14 continuous days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the trial vaccine. An immunosuppressant dose of glucocorticoid will be defined as a systemic dose ≥ 10 mg of prednisone per day or equivalent. The use of topical, inhaled, and nasal glucocorticoids will be permitted.
8. Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the trial vaccine.
9. Acute disease at the time of enrollment (defined as the presence of a moderate or severe illness with or without fever, or an oral temperature ≥ 38.0°C, on the planned day of vaccine administration).
10. Any condition that in the opinion of the investigator would pose a health risk to the subject if enrolled or could interfere with evaluation of the vaccine or interpretation of trial results (including neurologic or psychiatric conditions deemed likely to impair the quality of safety reporting).
11. Known disturbance of coagulation.
12. Suspicion or recent history (within 1 year of planned vaccination) of alcohol or other substance abuse.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 2654 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2020-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Novavax, Inc.
Locations (19):
- United States (19):
  - US135, Hollywood, Florida
  - US045, Savannah, Georgia
  - US013, Stockbridge, Georgia
  - US012, Meridian, Idaho
  - US032, Nampa, Idaho
  - US003, Lenexa, Kansas
  - US138, Rockville, Maryland
  - US025, Norfolk, Nebraska
  - US018, Omaha, Nebraska
  - US056, Binghamton, New York
  - US017, Endwell, New York
  - US030, Cleveland, Ohio
  - US053, Oklahoma City, Oklahoma
  - US044, Warwick, Rhode Island
  - US079, Mt. Pleasant, South Carolina
  - US050, Dakota Dunes, South Dakota
  - US029, Nashville, Tennessee
  - US004, San Antonio, Texas
  - US073, Tomball, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shinde V, Cho I, Plested JS, Agrawal S, Fiske J, Cai R, Zhou H, Pham X, Zhu M, Cloney-Clark S, Wang N, Zhou B, Lewis M, Price-Abbott P, Patel N, Massare MJ, Smith G, Keech C, Fries L, Glenn GM. Comparison of the safety and immunogenicity of a novel Matrix-M-adjuvanted nanoparticle influenza vaccine with a quadrivalent seasonal influenza vaccine in older adults: a phase 3 randomised controlled trial. Lancet Infect Dis. 2022 Jan;22(1):73-84. doi: 10.1016/S1473-3099(21)00192-4. Epub 2021 Sep 23. PMID 34563277

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NanoFlu | Fluzone Quadrivalent
Started | 1332 | 1322
Safety Population (The Safety Population was analyzed as actually treated (ie, based on the actual dose received).) | 1333 | 1319
Completed | 1312 | 1302
Not Completed | 20 | 20
Not completed — Lost to Follow-up | 11 | 8
Not completed — Adverse Event | 4 | 5
Not completed — Voluntary withdrawal unrelated to adverse event | 1 | 2
Not completed — Miscellaneous | 4 | 5

BASELINE CHARACTERISTICS:
Population: 2654 participants were randomized at a 1:1 ratio into 1 of 2 vaccine groups. Both groups were stratified by site, age (65 to < 75 and ≥ 75 years), and history of prior year receipt of the 2018-2019 influenza vaccine. The Safety Population was analyzed as actually treated (ie, based on the actual dose received).
Groups:
- Total: Total of all reporting groups
Arm/Group | NanoFlu | Fluzone Quadrivalent | Total
Number analyzed (Participants) | 1333 | 1319 | 2652
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.5 (5.7) | 72.5 (5.7) | 72.5 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 792 | 845 | 1637
  Male | 541 | 474 | 1015
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 64 | 65 | 129
  Not Hispanic or Latino | 1269 | 1254 | 2523
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 14 | 3 | 17
  Asian | 6 | 11 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 105 | 103 | 208
  White | 1208 | 1200 | 2408
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Received 2018-2019 Influenza Vaccine [Count of Participants; unit: Participants] | 1117 | 1102 | 2219
Received any influenza vaccination within the past 3 years [Count of Participants; unit: Participants] | 1210 | 1200 | 2410
Reaction from vaccine within the past 3 years [Count of Participants; unit: Participants] | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: HAI Antibody Responses for Vaccine Homologous Influenza Strains Expressed as Ratio of Geometric Mean Fold Ratio (GMFR)
Description: Egg-Based HAI Assay responses for all 4 vaccine homologous influenza strains (ie, 2 influenza A and 2 influenza B strains) expressed as GMFR on Day 28
Time Frame: Day 28
Population: Per-Protocol (PP) Population including all subjects who provided consent, were randomized and received the assigned dose of the test article according to protocol.
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Fold Ratio
Arm/Group | NanoFlu | Fluzone Quadrivalent
Number analyzed (Participants) | 1280 | 1286
Geometric Mean Fold Ratio
  A/Brisbane/02/2018 (H1N1) | 1.9 [1.8 to 2.0] | 1.7 [1. to 1.8]
  A/Kansas/14/2017 (H3N2) | 2.7 [2.6 to 2.9] | 2.3 [2.2 to 2.4]
  B/Maryland/15/2016 (Victoria lineage) | 1.6 [1.5 to 1.6] | 1.5 [1.5 to 1.6]
  B/Phuket/3073/2013 (Yamagata lineage) | 2.4 [2.3 to 2.5] | 2.0 [1.9 to 2.1]

2. Primary Outcome: Mean Difference in the Seroconversion Rate (SCR) HAI Antibody Responses for Vaccine Homologous Influenza Strains Expressed as a Percentage of Participants
Description: Egg-Based HAI Assay responses for all 4 vaccine homologous influenza strains (ie, 2 influenza A and 2 influenza B strains) summarized in terms of SCR on Day 28
Time Frame: Day 0 - Day 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NanoFlu | Fluzone Quadrivalent
Number analyzed (Participants) | 1280 | 1286
percentage of participants
  A/Brisbane/02/2018 (H1N1) pdm09 | 22.0 [19.8 to 24.4] | 17.0 [15.0 to 19.2]
  A/Kansas/14/2017 (H3N2) | 41.8 [39.1 to 44.6] | 34.4 [31.8 to 37.1]
  B/Maryland/15/2016 (Victoria lineage) | 11.2 [9.5 to 13.0] | 10.7 [9.0 to 12.5]
  B/Phuket/3073/2013 (Yamagata lineage) | 31.3 [28.8 to 33.9] | 22.9 [20.6 to 25.3]

3. Primary Outcome: Number of Subjects With Solicited Local and Systemic Adverse Events (AEs)
Description: Number of subjects with solicited local and systemic AEs over 7 days post-injection (ie, Day 0 through Day 6, inclusive).
Time Frame: Day 0 - Day 6
Population: Safety Population, including all study subjects who provided consent, were randomized, and received a test article. The Safety Population was analyzed as actually treated (ie, based on the actual dose received).
Measure: Number; unit: participants
Arm/Group | NanoFlu | Fluzone Quadrivalent
Number analyzed (Participants) | 1333 | 1319
participants
  Local solicited TEAEs | 372 | 243
  Systemic Solicited TEAEs | 369 | 292

4. Primary Outcome: Number of Subjects With Medically Attended Adverse Events (MAAEs), Serious Adverse Events (SAEs), Significant New Medical Conditions (SNMCs)
Description: Number of subjects with Medically Attended Adverse Events (MAAEs), Serious Adverse Events (SAEs), Significant New Medical Conditions (SNMCs) - including AESIs - through 1-year post-injection.
Time Frame: Day 0 - Day 364
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | NanoFlu | Fluzone Quadrivalent
Number analyzed (Participants) | 1333 | 1319
participants
  SAEs | 81 | 78
  SNMCs | 42 | 49
  MAAEs | 353 | 354

5. Primary Outcome: Number of Subjects With MAAEs, SAEs, SNMCs
Description: Number of subjects with MAEs, SAEs, and SNMCs - including AESIs.
Time Frame: Day 0 - Day 27
Population: Safety Population, including all study subjects who provided consent, were randomized and received a test article. The Safety Population was analyzed as actually treated (ie, based on the actual dose received).
Measure: Number; unit: participants
Arm/Group | NanoFlu | Fluzone Quadrivalent
Number analyzed (Participants) | 1333 | 1319
participants
  SAEs | 10 | 5
  SNMCs | 4 | 11
  MAAEs | 108 | 108

6. Secondary Outcome: HAI Titers to All Vaccine Homologous Influenza Strains and at Least 1 Antigenically Drifted Strain Expressed as Geometric Mean Titers (GMT)
Description: Homologous influenza strains and 1 antigenically drifted strain expressed as GMT
Time Frame: Day 0 - Day 28
Population: Per-Protocol (PP) Population including all subjects provided consent, were randomized and received the assigned dose of the test article according to protocol, had HAI serology results for Day 0 and Day 28, and had no major protocol deviations affecting the primary immunogenicity outcomes as determined by the sponsor prior to database lock and unblinding.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | NanoFlu | Fluzone Quadrivalent
Number analyzed (Participants) | 1280 | 1286
titers
  Day 0 - A/ Brisbane (H1N1) | 26.2 [25.0 to 27.4] | 26.0 [24.9 to 27.1]
  Day 28 - A / Brisbane (H1N1) | 49.3 [46.7 to 51.9] | 45.0 [42.7 to 47.3]
  Day 0 - A/ Kansas (H3N2) | 55.1 [53.5 to 56.8] | 54.7 [53.1 to 56.3]
  Day 28- A/ Kansas (H3N2) | 151.5 [143.3 to 160.2] | 126.8 [120.3 to 133.6]
  Day 0 - B (Victoria Lineage) | 70.7 [68.0 to 73.5] | 69.8 [67.2 to 72.5]
  Day 28 - B (Victoria Lineage) | 110.7 [106.1 to 115.6] | 106.3 [102.3 to 110.6]
  Day 0 - B (Yamagata Lineage) | 69.1 [66.0 to 72.3] | 66.5 [63.6 to 69.6]
  Day 28- B (Yamagata Lineage) | 168.5 [160.2 to 177.2] | 133.9 [127.7 to 140.5]
  Day 0 - A/California (H3N2) | 44.5 [42.4 to 46.7] | 44.0 [42.0 to 46.0]
  Day 28- A/California (H3N2) | 115.0 [108.0 to 122.4] | 80.6 [75.9 to 85.6]

7. Secondary Outcome: HAI Titers to All Vaccine Homologous Influenza Strains and at Least 1 Antigenically Drifted Strain Expressed as Geometric Mean Fold Ratio (GMFR)
Description: Wild-Type HAI Assay Homologous influenza strains and 1 antigenically drifted strain expressed as GMFR.
Time Frame: Day 28 - 364
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Fold Rise
Arm/Group | NanoFlu | Fluzone Quadrivalent
Number analyzed (Participants) | 1280 | 1286
Geometric Mean Fold Rise
  Day 28- A/Brisbane (H1N1) | 2.4 [2.3 to 2.5] | 1.9 [1.8 to 2.0]
  Day 28 - A/Kansas (H3N2) | 5.6 [5.3 to 6.0] | 3.4 [3.2 to 3.6]
  Day 28 - B/ Maryland (Victoria Lineage) | 2.1 [2.0 to 2.2] | 1.6 [1.5 to 1.7]
  Day 28 - B/Phuket (Yamagata Linage) | 2.6 [2.5 to 2.7] | 1.8 [1.7 to 1.8]
  Day 28 - A/California (H3N2) | 2.6 [2.5 to 2.7] | 1.8 [1.8 to 1.9]
  Day 28 - A/Cardiff (H3N2) | 2.4 [2.3 to 2.5] | 1.8 [1.7 to 1.8]
  Day 364- A/Brisbane (H1N1) | 2.0 [1.6 to 2.5] | 2.0 [1.6 to 2.4]
  Day 364 - A/Kansas (H3N2) | 2.9 [2.3 to 3.6] | 2.2 [1.9 to 2.7]
  Day 364 - B/ Maryland (Victoria Lineage) | 2.0 [1.7 to 2.2] | 1.8 [1.6 to 2.0]
  Day 364 - B/Phuket (Yamagata Linage) | 1.1 [1.0 to 1.3] | 1.1 [0.9 to 1.2]
  Day 364 - A/California (H3N2) | 79.6 [65.8 to 96.2] | 75.7 [65.5 to 87.3]
  Day 364 - A/Cardiff (H3N2) | 2.0 [1.7 to 2.4] | 1.5 [1.2 to 1.7]

8. Secondary Outcome: Subjects Who Seroconverted as Determined by HAI Titers to All Vaccine Homologous Influenza Strains and at Least 1 Antigenically Drifted Strain
Description: Wild-Type HAI Assay Homologous Influenza Strains and at least 1 Antigenically Drifted Strain Expressed as Seroconversion Rate (SCR).
Time Frame: Day 28 - Day 364
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NanoFlu | Fluzone Quadrivalent
Number analyzed (Participants) | 1280 | 1286
percentage of participants
  Day 28- A/Brisbane/02/2018 (H1N1) pdm09 | 32.7 [30.2 to 35.4] | 21.4 [19.2 to 23.7]
  Day 28-A/Kansas/14/2017 (H3N2) | 69.8 [67.2 to 72.3] | 49.5 [46.7 to 52.2]
  Day 28- B/Maryland/15/2016 (Victoria lineage) | 25.1 [22.7 to 27.5] | 13.5 [11.6 to 15.4]
  Day 28- B/Phuket/3073/2013 (Yamagata lineage) | 35.4 [32.8 to 38.1] | 17.7 [15.7 to 19.9]
  Day 28 - A/California (H3N2) | 37.1 [34.5 to 39.8] | 20.5 [18.4 to 22.8]
  Day 28 - A/Cardiff (H3N2) | 32.7 [30.2 to 35.4] | 18.6 [16.5 to 20.8]
  Day 364 - A/California (H3N2) | 19.0 [10.2 to 30.9] | 5.4 [1.1 to 14.9]
  Day 364 - A/Cardiff (H3N2) | 22.2 [12.7 to 34.5] | 7.1 [2.0 to 17.3]
  Day 364- A/Brisbane/02/2018 (H1N1) pdm09 | 19.0 [10.2 to 30.9] | 19.6 [10.2 to 32.4]
  Day 364-A/Kansas/14/2017 (H3N2) | 54.0 [40.9 to 66.6] | 28.6 [17.3 to 42.2]
  Day 364- B/Maryland/15/2016 (Victoria lineage) | 17.5 [9.1 to 29.1] | 8.9 [3.0 to 19.6]
  Day 364- B/Phuket/3073/2013 (Yamagata lineage) | 6.3 [1.8 to 15.5] | 3.6 [0.4 to 12.3]

9. Secondary Outcome: Subjects Who Seroprotected as Determined by HAI Titers to All Vaccine Homologous Influenza Strains and at Least 1 Antigenically Drifted Strain Expressed as SPR
Description: Homologous Influenza Strains and at least 1 Antigenically Drifted Strain Expressed as Seroprotection Rate (SPR).
Time Frame: Day 28
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NanoFlu | Fluzone Quadrivalent
Number analyzed (Participants) | 1280 | 1286
percentage of participants
  A/Brisbane/02/2018 (H1N1) pdm09 | 69.1 [66.4 to 71.6] | 64.5 [61.9 to 67.2]
  A/Kansas/14/2017 (H3N2) | 98.8 [98.1 to 99.3] | 98.3 [97.4 to 98.9]
  B/Maryland/15/2016 (Victoria lineage) | 99.1 [98.5 to 99.6] | 98.7 [97.9 to 99.2]
  B/Phuket/3073/2013 (Yamagata lineage) | 99.0 [98.6 to 99.5] | 97.5 [96.5 to 98.3]

ADVERSE EVENTS:
Time Frame: 1 year
Description: Serious Adverse Events
Arm/Group | NanoFlu | Fluzone Quadrivalent
All-Cause Mortality (participants affected / at risk) | 8/1333 | 8/1319
Serious Adverse Events (participants affected / at risk) | 136/1333 | 125/1319
Other Adverse Events (participants affected / at risk) | 0/1333 | 0/1319
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NanoFlu (N=1333) | Fluzone Quadrivalent (N=1319)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 3 (3)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 4 (4) | 4 (4)
Coronary artery disease (Cardiac disorders) | 3 (3) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocutaneous fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 4 (4)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Complication associated with device (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Ischaemic hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 3 (3)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 4 (4) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis staphylococcal (Infections and infestations) | 2 (2) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (2) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Localised infection (Infections and infestations) | 3 (3) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 1 (1)
Pelvic abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 8 (8) | 6 (6)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1)
Postoperative abscess (Infections and infestations) | 0 (0) | 1 (1)
Renal abscess (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 4 (4) | 2 (2)
Septic shock (Infections and infestations) | 1 (1) | 1 (2)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hormone receptor positive breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery disease (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 2 (2)
Transient aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Transient global amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 2 (2)
Anuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Accelerated hypertension (Vascular disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Arterial spasm (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive urgency (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/94/NCT04120194/Prot_002.pdf
  • Statistical Analysis Plan (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT04120194/SAP_001.pdf